CLINICAL TRIAL: NCT01731366
Title: Gut, Grain and Greens (3G): The Effect of Wholegrain on Gut Microbiome and Metabolic Health
Brief Title: The Effect of Whole Grain on Gut Microbiome and Metabolic Health
Acronym: 3G
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: Technical University of Denmark (Other)
Responsible Party: Principal Investigator, Arne Astrup, Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: M206
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Metabolic Disease; Injury of Gastrointestinal Tract
MeSH Terms: conditions — Metabolic Diseases | interventions — Whole Grains

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Refined grain (Placebo Comparator): Refined grain diet: Participants consume less than 10 g of whole grain per day (corresponds to the whole grain intake below the 10th percentile of the population)
  Interventions: Other: Refined grain
- Whole grain (Active Comparator): Whole grain diet: Participants consume more than 75g of whole grain per day (corresponds to the whole grain intake of the 90th percentile of the population)
  Interventions: Other: Whole grain

INTERVENTIONS:
Other: Whole grain — Whole grain diet: Participants consume more than 75g of whole grain per day (corresponds to the whole grain intake of the 90th percentile of the population)
  Arms: Whole grain
Other: Refined grain — Refined grain diet: Participants consume less than 10 g of whole grain per day (corresponds to the whole grain intake below the 10th percentile of the population)
  Arms: Refined grain

SUMMARY:
Objective: To identify how specific changes of the whole grain content in the diet affect the host-gut microbiome interactions with implications for metabolic health .

Design: A randomized, controlled, single-blinded, cross-over intervention trial consisting of two 8-week intervention periods, separated by a 6-week wash-out period. A total of 60 participants will be included.

Intervention: low vs. high whole grain intake.

DETAILED DESCRIPTION:
The study is designed as a randomized, controlled, single-blinded, cross-over intervention trial consisting of two 8-week interventions periods, separated by a 6-week wash-out period. A total number of 60 participants will be included. Participants consume, in randomized order, a diet rich in whole grain in the active treatment period and a refined grain diet during the control period.

Measurements: Insulin sensitivity will be assessed by means of a meal challenge test and by the Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) which is the primary outcome of this study. Secondary outcomes include metabolic and inflammatory markers, appetite hormones, transit time, and GM composition. Furthermore, selected control measures are included; 4-day food records and a study intervention diary.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI): 25 - 35 kg/m2
* No medical prescribed diet
* Weight stable
* No blood donation during the study
* Intense sporting activities less than 10h/ week
* Alcohol consumption less than 14 units/ week (female) and 21 units/ week (male)
* Signed written consent

Exclusion Criteria:

* Pharmacological treatment; hypertension, diabetes and blood lipid regulation
* Lactating (or lactating, 6 weeks ago), pregnant (or pregnant, 3 months ago) or wish to become pregnant during the study
* Participation in another biomedical trial 1 month prior to study start
* Diagnosed with any form of diabetes, celiac disease or chronic pancreatitis
* Reported chronic gastrointestinal disorders
* Antibiotic treatment for 3 month prior to study start
* Intake of vitamin, mineral, or pre- or probiotic supplements for 1 month prior to study start
* Blood hemoglobin < 7.0 mmol/l
* Blood donation within 1 month prior to study start

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-02 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
HOMA-IR | At the end of the intervention periods
  Homeostasis Model Assessment of fasting Insulin Resistance (HOMA-IR: glucose (mmol/l( x insulin (pmol/l)/22.5)
Metagenomic profile | At the end of the intervention periods
  Altered quantitative metagenomics at bacterial gene- and species levels, which is a non-specific outcome, but included as the main hypothesis of the project is to test if HOMA-IR is affected via changes in the gut microbiome.

SECONDARY OUTCOMES:
Mean intestinal transit time | At the end of the intervention periods
  Participants are instructed in swallowing capsules containing different small non-invasive and non-absorbable plastic pellets for 6 consecutive days. On the seventh day they are having an X-ray of the abdomen taken.
Gastrointestinal permeability, Lactulose/ mannitol ratio | At the end of the intervention periods
  5 hours urine collection following intake of lactulose and mannitol
Colonic fermentation | At the end of the intervention periods
  Measurement of breath hydrogen excretion (at before and 30, 60, 90, 120, 150, 180 after intake of standard breakfast) and plasma short-chain fatty acids (fasting and 30, 60, 120, 180 minutes after standard breakfast)
Saliva microbial flora | At the end of the intervention periods
  Determination of fasting microbial composition of flora.
Blood pressure | At the end of the intervention periods
  Measurement of supine systolic and diastolic blood pressure (3 times)
Appetite hormones | At the end of the intervention periods
  Determination of different appetite hormones in fasting and postprandial blood samples (30, 60, 120, 180 minutes after standard breakfast)
Blood lipid profile | At the end of the interventions periods
  Measurement of different blood lipids in fasting and postprandial blood samples (30, 60, 120, 180 minutes after standard breakfast)
Body composition | At the end of the intervention periods
  Measurement of body fat mass and percentage via bio-impedance
Subjective appetite sensation | At the end of the intervention periods
  Assessment of subjective appetite sensation via visual analogue scales
Energy intake | At the end of the intervention periods
  Assessment of energy intake at an ad libitum meal 3 hours after a standard breakfast
Ex vivo cytokine production | At the end of the intervention periods
  Production of cytokines (such as IL-1beta, IL-6) in stimulated whole blood cultures.
Gene expression | At the end of the intervention periods
  Assessed by mRNA qPCR in whole blood and cells from whole blood stimulation. Main focus is put on genes involved in immune function and metabolic regulation.
Immune cell profiling | At the end of the intervention periods
  Assessed by flow cytometry of whole blood.
Immune markers | At the end of the intervention periods
  Fasting plasma cytokines, hsCRP, and LPS/LPS-BP
Blood immune cell content | At the end of the intervention periods
  Assessed by hematological cell counts
Markers og glucose hemostasis | At the end of the intervention periods
  Measurement of plasma concentrations of Insulin, Proinsulin and HbA1c
Markers of one-carbon metabolism | At the end of the intervention periods
  Assessed by plasma homocystein, SAM/SAH and betain
Plasma adipokines | December 2015
  Leptin and adiponectin

OTHER OUTCOMES:
4-days precoded food diary | December 2014
  Assessment of dietary intake via food frequency questionnaire as a measure of compliance
n-3 fatty acid status | At the end of the intervention periods
  Assessed as DHA percentage in a whole blood fatty acid analysis. Included as a potential effect modificator in relation to immune function and metabolic outcomes.
Alkyresorcinol | At the end of the intervention periods
  Measured in plasma as a marker of compliance to the whole grain intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Lotte Lauritzen, Associate professor, Principal Investigator — University of Copenhagen
Locations (1):
- Department of Human Nutrition, University of Copenhagen, Fredriksberg, Denmark

REFERENCES:
- [Derived] Lind MV, Lauritzen L, Vestergaard H, Hansen T, Pedersen O, Kristensen M, Ross AB. One-carbon metabolism markers are associated with cardiometabolic risk factors. Nutr Metab Cardiovasc Dis. 2018 Apr;28(4):402-410. doi: 10.1016/j.numecd.2018.01.005. Epub 2018 Jan 31. PMID 29499850
- [Derived] Roager HM, Vogt JK, Kristensen M, Hansen LBS, Ibrugger S, Maerkedahl RB, Bahl MI, Lind MV, Nielsen RL, Frokiaer H, Gobel RJ, Landberg R, Ross AB, Brix S, Holck J, Meyer AS, Sparholt MH, Christensen AF, Carvalho V, Hartmann B, Holst JJ, Rumessen JJ, Linneberg A, Sicheritz-Ponten T, Dalgaard MD, Blennow A, Frandsen HL, Villas-Boas S, Kristiansen K, Vestergaard H, Hansen T, Ekstrom CT, Ritz C, Nielsen HB, Pedersen OB, Gupta R, Lauritzen L, Licht TR. Whole grain-rich diet reduces body weight and systemic low-grade inflammation without inducing major changes of the gut microbiome: a randomised cross-over trial. Gut. 2019 Jan;68(1):83-93. doi: 10.1136/gutjnl-2017-314786. Epub 2017 Nov 1. PMID 29097438
- [Derived] Lind MV, Madsen ML, Rumessen JJ, Vestergaard H, Gobel RJ, Hansen T, Lauritzen L, Pedersen OB, Kristensen M, Ross AB. Plasma Alkylresorcinols Reflect Gluten Intake and Distinguish between Gluten-Rich and Gluten-Poor Diets in a Population at Risk of Metabolic Syndrome. J Nutr. 2016 Oct;146(10):1991-1998. doi: 10.3945/jn.116.236398. Epub 2016 Sep 14. PMID 27629576
- See also: Related Info — http://www.3g-center.dk/